CLINICAL TRIAL: NCT06006780
Title: Porcine Acellular Dermal Matrix for the Treatment of Localized Gingival Recessions: A Multicenter Randomized Clinical Trial
Brief Title: Porcine Acellular Dermal Matrix for the Treatment of Localized Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Enilson Antonio Sallum, PhD, Chair of Periodontolgy Area, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 59036822.4.1001.5418
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coronally advanced flap (CAF) (Active Comparator)
  Interventions: Other: Coronally advanced flap (CAF)
- Coronally advanced flap associated with the porcine acellular dermal matrix (CAF+ PADM) (Experimental)
  Interventions: Device: Porcine acellular dermal matrix

INTERVENTIONS:
Device: Porcine acellular dermal matrix — Coronally advanced flap associated with the porcine acellular dermal matrix for root coverage
  Other Names: Mucoderm
  Arms: Coronally advanced flap associated with the porcine acellular dermal matrix (CAF+ PADM)
Other: Coronally advanced flap (CAF) — Coronally advanced flap for root coverage
  Arms: Coronally advanced flap (CAF)

SUMMARY:
Aim: The aim of this randomized clinical trial is to evaluate the use of the porcine acellular dermal matrix (PADM) for the treatment of RT1 localized gingival recessions.

Material and methods: Forthy patients (n=20) with RT1 localized gingival recessions with height ranging from 3 to 5 mm with and at least, 2mm of keratinized tissue width will be selected to participate in the study. Patients will be allocated randomly in two treatment groups: Coronally advanced flap (CAF) or coronally advanced flap associated with the porcine acellular dermal matrix (CAF+ PADM). The clinical parameters evaluated at the baseline, 6 and 12 months will be: Plaque index (IPL); gingival index (GI); relative gingival recession height (RGRH); gingival recession width (GRW); probing depth (PD); relative clinical attachment level (RCAL); keratinized tissue height (KTH); keratinized tissue thickness (KTT); papilla height (PH). Evaluations will be made by the professional and the patient regarding dentin hypersensitivity (HD) (Schiff and VAS scales respectively), aesthetics (RES and VAS scales, respectively) and patient's centered outcomes, through the questionnaire referring to the OHIP-14.

Descriptive statistical analysis will be expressed as mean ± standard deviation (SD), median, quartiles, percentages and confidence intervals (95% CI). To analyze the normality of the residue, the Shapiro-Wilk test will be performed. Then, the Wilcoxon test will be applied to compare the periodontal parameters and a quality of life, before and post-treatment. Correlations between parameters and dental hypersensitivity will be analyzed through Spearman's test. Key words: Gingival recession, Root coverage, Biomaterial, Acellular dermal matrix.

ELIGIBILITY:
Inclusion Criteria:

* RT1 localized gingival recessions with height ranging from 3 to 5 mm;
* 2mm or more of keratinized tissue width ;
* Probing depth less than 3mm;
* Plaque and gingival index less or equal to 20%.

Exclusion Criteria:

* Smokers;
* Pregnants;
* Nursing;
* Patients with diabetes mellitus or another condition that interfere in the tissue repair
* Patients who use drugs or medications that interfere in the tissue repair;
* Allergies to any composition of the devices of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Recession change | Baseline, 6 months and 12 months
  Change of the gingival recession height

SECONDARY OUTCOMES:
Thickness of keratinized tissue | Baseline, 6 months and 12 months
  Thickness of keratinized tissue evaluation after periodontal plastic surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Piracicaba Dental School, State University of Campinas, Piracicaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sangiorgio JPM, Neves FLDS, Rocha Dos Santos M, Franca-Grohmann IL, Casarin RCV, Casati MZ, Santamaria MP, Sallum EA. Xenogenous Collagen Matrix and/or Enamel Matrix Derivative for Treatment of Localized Gingival Recessions: A Randomized Clinical Trial. Part I: Clinical Outcomes. J Periodontol. 2017 Dec;88(12):1309-1318. doi: 10.1902/jop.2017.170126. Epub 2017 Jul 28. PMID 28753100